CLINICAL TRIAL: NCT06179602
Title: Prospective Cohort Study on Thermal Ablation of Malignant Liver Tumors Within the IMAGIO Project (A-IMAGIO)
Brief Title: Prospective Cohort Study on Thermal Ablation of Malignant Liver Tumors
Acronym: A-IMAGIO
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Philips Healthcare (Industry); European Commission (Other)
Responsible Party: Principal Investigator, Mark C Burgmans, MD PhD, Dr. M. C. Burgmans, MD PhD, Leiden University Medical Center
Other Study IDs: 133356
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-09

CONDITIONS: Liver Cancer; Liver Metastases; Liver Metastasis Colon Cancer; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The endpoint of this study is to develop and validate algorithms, using artificial intelligence and machine learning, to optimize patient selection, treatment planning, treatment evaluation and outcome prediction in patients undergoing thermal ablation of a malignant liver tumor. The long-term objective is to establish thermal ablation as the treatment of choice for the vast majority of patients with a primary or secondary liver tumor by development of an accessible workflow that can be widely implemented in different centers performing thermal ablation. Over a time span of at least four years, data will be collected prospectively, encompassing patient information, tumor characteristics, and treatment details. Additionally, pre-, intra-, and post-procedural imaging will be systematically gathered.

DETAILED DESCRIPTION:
This study is part of the IMAGIO (Imaging and advanced guidance for workflow optimization in interventional oncology) project. This project aims to leverage Interventional Oncology in the clinical setting to improve cancer survival outcomes, through minimally invasive, efficient and affordable care pathways for three disease states; liver cancer, lung cancer and sarcoma. In IMAGIO, top innovators in MedTech and Pharma and expert academic clinical centers will mature the next-generation interventional oncology imaging across the full spectrum, from pre-clinical developments to impact validation in clinical trials.

The objective of this study, A-IMAGIO, is to develop a standardized, accessible, low-complex, end-to-end solution for patient selection, treatment planning, needle guidance and treatment evaluation for thermal liver ablation.

One of the objectives is to integrate AI in the clinical workflow as a tool to assist operators in decision making throughout the entire process based on quantitative assessment. AI data analytics will be developed to guide decision making for personalized treatment together with algorithms that allow optimized treatment planning and automated quantitative treatment evaluation. Also, a computational model will be developed with input from radiomics and clinical data to identify patients at risk of recurrence after thermal ablation. The aim of the A-IMAGIO project is to conduct a large European observational cohort study and collect clinical and image data of patients treated with thermal ablation for liver tumors in order to develop and validate these AI algorithms. The database will be built by merging data from retrospective data and previous prospective clinical trials on thermal ablation of liver tumors. Further data will be collected through a prospective, multicenter, observational study. The long-term objective is to establish thermal ablation as the first line therapy for patients with both primary and secondary liver tumors. Therefore, we aim to develop a low-complexity-high-precision, accessible workflow that can be widely implemented in different centers performing thermal ablation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above
* Candidate for percutaneous thermal liver ablation as discussed in a multidisciplinary tumorboard (MDT)
* Informed consent

Exclusion Criteria:

* Patients lacking capacity to give informed consent.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with one or more primary or secondary liver malignancy who are candidates for thermal liver ablation as discussed in a multidisciplinary tumour board.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy as assessed by local recurrence | Throughout the entire four-year study period
Efficacy as assessed by time-to-recurrence | Throughout the entire four-year study period
Efficacy as assessed by disease-free-survival | Throughout the entire four-year study period
Efficacy as assessed by overall survival | Throughout the entire four-year study period
Safety as assessed by complications according to CTCAE v6.0. | Throughout the entire four-year study period
  Treatment related adverse events are defined as grade 3-4 adverse events and serious

CONTACTS AND LOCATIONS:
Overall Officials: Mark C. Burgmans, MD PhD, Principal Investigator — Leiden univeristy medical centre; Christiaan van der Leij, MD PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van der Velden AL, Verhagen CAM, Gholamiankhah F, Rahmani H, van Dam RM, van Duijn-de Vreugd JJ, Simon SR, Hendriks P, van Erp GCM, Knapen RRMM, Volmer L, Overduin K, Braak JPBM, Bale R, Laimer G, Lanocita R, Meijerink MR, Kampfer Y, Denys A, Littler P, Sternberg B, Kobeiter H, Smits MLJ, van Strijen MJL, Pieterman KJ, Broersen A, Dijkstra J, Brecheisen R, Burgmans MC, van der Leij C. Prospective Registry Study on Thermal Liver Ablation of Primary and Secondary Liver Tumours Named the A-IMAGIO Study. Cardiovasc Intervent Radiol. 2025 Aug;48(8):1193-1199. doi: 10.1007/s00270-025-04093-9. Epub 2025 Jun 23. PMID 40550852